CLINICAL TRIAL: NCT04517513
Title: Shanghai Community Cohort Establishment and Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Jinqiao Community Health Service Center of Pudong new area, Shanghai (Unknown); Heqing Community Health Service Center of Pudong new area, Shanghai (Unknown); Weifang Community Health Service Center of Pudong new area, Shanghai (Unknown); Jinyang Community Health Service Center of Pudong new area, Shanghai (Unknown)
Responsible Party: Principal Investigator, Jun Pu, Director of Cardiovascular Medicine, RenJi Hospital
Other Study IDs: Shanghai Community Cohort
Record Dates: First submitted 2020-08-16; First posted 2020-08-18 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Diseases
Keywords: Cohort Study; Natural Population; China
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Biological specimen collection: collect 10ml ethylenediaminetetraacetic acid blood samples using a health checkup, then send them to renji sample bank for separation within 2 hours, and store in -80℃ ultra-low temperature refrigerator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective is to establish a natural population cohort in East China based on the latest scientific researches, preliminary findings of the project team, and a close cooperation model of the Specialist Medical Consortium.

Firstly, we will focus on the information and management status of high-risk, single-patient, and co-occurring patient groups of cardio cerebral diseases such as coronary heart disease and stroke. We plan to integrate the questionnaire data and sample database information into the cardio-cerebral "co-prevention and management" information platform, in order to establish a cardiovascular and cerebrovascular disease management system.

Secondly, we aim to develop a new risk prediction model for heart and brain diseases based on the big data platform, lead the establishment of the "co-prevention and management" innovation management model for cardio cerebral diseases, and explore an integrated and innovative health management model for the prevention and treatment of cardio cerebral diseases for China.

DETAILED DESCRIPTION:
The research is based on a combination of retrospective, cross-sectional, and prospective cohort studies.

In particular, the retrospective cohort study collects historical information of the studied cohort from 2014 to 2018 from secondary medical units, residents' community health service centers, emergency departments, and their health records. Patients' past diseases such as hypertension, diabetes, cardiovascular and cerebrovascular diseases, information on the history of drug use, and lifestyle (if any) are collected and sorted out. Moreover, information on cardiovascular and cerebrovascular morbidity and death among members of the cohort is collected.

The cross-sectional study builds on the baseline research conducts during 2019-2020. Specifically, baseline research contains the following procedures:

1. Epidemiological survey: Design the Cardio-Cerebrovascular Disease Prevention and Control Questionnaire in accordance with the principles and requirements of the cohort study. On the premise of informed notification, data are collected through face-to-face interviews between the studied cohort and investigators who signed the informed consent and received uniform training. Quality control staff will review the questionnaire for quality control. The main content includes demographic sociology, lifestyle, physical exercise, daily eating habits, usage of dietary supplements, personal and family medical history, psychological assessment, and female fertility history.
2. Physical examination: the examination is performed by the clinical professional physician in the health service center. The examination content includes height, weight, blood pressure, hearing, vision, internal surgery, body fat composition (optional), chest radiograph, electrocardiogram, B-ultrasound, carotid ultrasound (optional), and other imaging examinations.
3. Clinical biochemical test: fasting blood collection should be performed by all individuals upon their enrollment. The blood samples collected are tested for biochemistry, liver and kidney function, blood lipid analysis, and electrolyte analysis in accordance with clinical testing requirements.
4. Biological specimen collection: collect 10ml ethylenediaminetetraacetic acid blood samples using a health checkup, then send them to renji sample bank for separation within 2 hours, and store in -80℃ ultra-low temperature refrigerator.

Lastly, the prospective study will be conducted from 2020 to 2025. Through annual active (phone, face-to-face interview, etc.) and passive follow-ups, we track the health status of the cohort including cardio-cerebral vascular disease occurrence, death, migration, etc., collect data that matches its baseline value, analyze the morbidity and mortality of the cohort population, and grasp the morbidity, the order of the diseases, mortality, and order of the cause of death for each disease, especially the cardiovascular and cerebrovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 35y
* Registered Permanent residents or have lived for more than 5 years and have local social security medical insurance
* Patients with no serious physical disability and can communicate normally
* Patients who participate voluntarily and sign informed consent
* Patients whose diseases and deaths are managed by the local health department

Exclusion Criteria:

* Temporary residents and floating population
* Patients with serious health conditions and cannot participate in the investigation
* Patients who are unwilling to accept follow-up inspections of the project

Min Age: 35 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible residents from second-class medical units and community health service centers with mature conditions.
Sampling Method: Non-Probability Sample
Enrollment: 80000 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular and Cerebrovascular incidence | 5 years
  Incidence of Cardiovascular and Cerebrovascular disease were calculated by age, gender and area compared by different health management mode.
Cardiovascular and Cerebrovascular mortality | 5 years
  Mortality of Cardiovascular and Cerebrovascular disease were calculated by age, gender and area compared by different health management mode.

SECONDARY OUTCOMES:
Normalized management rate of Cardiovascular and Cerebrovascular disease | 5 years
  Normalized management rate of Cardiovascular and Cerebrovascular disease were calculated by different management mode.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD,PhD, Principal Investigator — RenJi Hospital
Locations (1):
- Ren Ji Hospital Afflited to School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China